CLINICAL TRIAL: NCT06159634
Title: Comparison of the Efficacy of Using a Traction Device in Colonic Endoscopic Submucosal Dissection Versus Conventional ESD: A Randomized Clinical Trial
Brief Title: Traction vs. No Traction in Colonic ESD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Micro-Tech Endoscopy USA (Unknown)
Responsible Party: Principal Investigator, Mohamed Othman, MD, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-53522
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Gastrointestinal Neoplasm
Keywords: Endoscopic Submucosal Dissection; Endoscopic Traction
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into one of two arms: Conventional ESD, or ESD with traction device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ESD with traction device (Experimental): ESD of target lesion will be performed with the assistance of a traction device.
  Interventions: Procedure: Endoscopic Submucosal Dissection; Device: Traction Device
- Control arm (Active Comparator): ESD of target lesion will be performed without the use of a traction device
  Interventions: Procedure: Endoscopic Submucosal Dissection

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection — Endoscopic submucosal dissection (ESD) will be the technique used to remove target lesions.
Device: Traction Device — Use of traction device to aid in removing target lesions
  Arms: ESD with traction device

SUMMARY:
The goal of this prospective, randomized, controlled trial conducted at Baylor St. Luke's Medical Center is to compare the effectiveness and clinical outcomes of using a traction device in colonic endoscopic submucosal dissection (ESD) to those of using conventional ESD.

The investigators of this study hypothesize that use of the traction device will help expedite colonic endoscopic submucosal dissections.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is the mainstay for the treatment of complex colorectal polyps particularly those with a higher risk of superficial submucosal invasion. However, colonic ESD is technically difficult given the thin colon wall and difficult locations of lesion. Endoscopic submucosal dissection (ESD) of colonic lesions can be difficult because the thins wall of the colon wall and the lack of submucosal space expansion to the degree seen in the submucosal dissection in the esophagus or the stomach. ESD can be done in a standard fashion with circumferential incision followed by submucosal dissection according to gravity, tunneling methods, pocket methods or traction. Traction is frequently used to expedite submucosal dissection in particularly in tough locations or in fibrotic lesions. Traction assisted ESD is particularly attractive in colonic ESD given the above-mentioned difficulties and the challenge with performing other techniques such as tunneling or pocket formation in fibrotic lesions or lesions over folds. Tissue traction can be applied by several methods including gravity, mucosal tension, water pressure, and adjusting the patient's body position. Traction can also be applied using devices such as clip and line, snare or using additional endoscope. Data regarding the value of traction in colonic ESD is controversial. Despite multiple publications about the efficacy of traction devices in the east, there are few published data from the west. The Sure trac system was recently approved in the US for traction assisted ESD. The system has 2 devices, the primary device comes preloaded with a silicone band, while the secondary device features a clip of the same size as the primary device to apply traction on the opposite wall. Traction with sure trac system, is readily assembled and easily accessible and it is equipped with its own clip for swift implementation, thus expediting the process. The purpose of this research is to compare the effectiveness and safety of the sure trac traction system (Micro Tec endoscopy, USA) to standard ESD without applying traction.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years old.
2. Patients can provide informed consent.
3. Patient is referred for ESD procedure of colonic neoplastic lesions and with one of the following criteria:

A- Lesions with prior resection or with scar at any size. B- Granular lateral spreading tumors (GLST) more than 3 cm. C- Non granular lateral spreading tumors (NGLST) more than 20 mm. D- Any suspected submucosal invasion such as Paris classification II a +II or lesions with positive non lifting sign.

Exclusion Criteria:

1. Patient is < 18 years old.
2. Patient refused and/or unable to provide consent.
3. Patient is a pregnant woman.
4. Lesions with morphology: pedunculated type (Paris IP, Ips).
5. Appendiceal orifice or IC valve lesions. 6. Patients with lesions removed with other techniques besides ESD (like hybrid ESD or submucosal tunneling technique STER and EMR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dissection speed | Day 1 (procedure day)
  Length of time to perform endoscopic submucosal dissection by the operator as measured by calculating area of lesion divided by time (cm^2/hours).

SECONDARY OUTCOMES:
En-bloc, R0, and curative resection rates | Day 1 (procedure day)
  As collected for each group
Total procedure time | Day 1 (procedure day)
  Total procedure time to perform ESD from scope in to scope out
Intraprocedural adverse events | Day 1 (procedure day), up to 48 hours after procedure.
  Such as muscularis propria injury and bleeding (related to or not related to the traction devices).
Post-procedural adverse events | 1 month post-procedure
  As reported per subject follow-ups with the patient within 1 month.
Abdominal pain | 1 hour post-procedure, 24 hours post-procedure.
  Collected at 1 hour and 24 hours after procedure utilizing the Visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Othman, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - Baylor St. Lukes Medical Center (BSLMC), Houston, Texas

IPD SHARING:
Plan to Share IPD: No
There is no expected significant increased risk associated with the use of the traction device in ESD beyond what the current standard is for the procedure. Loss of confidentiality is the only other risk associated with this project. All measures to ensure patient confidentiality will be employed. Data will be coded and entered into a password-protected computer. Only the Principal Investigator and Study Research Coordinators will have access to data with patient identifiers. There will be no disclosure of a patients protected health information. Paper copies of the study documents will be created only as needed and only shown to the investigators listed in the study. Once the study is completed, all paper copies will be destroyed. If the results of the study are published or used in any presentations, all patient related information will be coded.

REFERENCES:
- [Background] Tanaka S, Terasaki M, Kanao H, Oka S, Chayama K. Current status and future perspectives of endoscopic submucosal dissection for colorectal tumors. Dig Endosc. 2012 May;24 Suppl 1:73-9. doi: 10.1111/j.1443-1661.2012.01252.x. PMID 22533757
- [Background] Othman MO, Jawaid SA, Rungta M, Sur N, Dhingra S. Double-balloon endolumenal intervention platform with flexible grasper to expedite colonic endoscopic submucosal dissection. VideoGIE. 2020 Dec 26;6(3):144-146. doi: 10.1016/j.vgie.2020.11.014. eCollection 2021 Mar. No abstract available. PMID 33738368
- [Background] Tamaru Y, Kuwai T, Miyakawa A, Kanazawa N, Kusunoki R, Shimura H, Uchiyama S, Ishaq S, Kohno H. Efficacy of a Traction Device for Endoscopic Submucosal Dissection Using a Scissor-Type Knife: A Randomized Controlled Trial. Am J Gastroenterol. 2022 Nov 1;117(11):1797-1804. doi: 10.14309/ajg.0000000000002019. Epub 2022 Sep 26. PMID 36191269
- [Background] Nagata M. Usefulness of underwater endoscopic submucosal dissection in saline solution with a monopolar knife for colorectal tumors (with videos). Gastrointest Endosc. 2018 May;87(5):1345-1353. doi: 10.1016/j.gie.2017.11.032. Epub 2017 Dec 12. PMID 29242059
- [Background] Yamasaki Y, Takeuchi Y, Uedo N, Kato M, Hamada K, Aoi K, Tonai Y, Matsuura N, Kanesaka T, Yamashina T, Akasaka T, Hanaoka N, Higashino K, Ishihara R, Iishi H. Traction-assisted colonic endoscopic submucosal dissection using clip and line: a feasibility study. Endosc Int Open. 2016 Jan;4(1):E51-5. doi: 10.1055/s-0041-107779. Epub 2015 Nov 30. PMID 26793785
- [Background] Burgess NG, Bassan MS, McLeod D, Williams SJ, Byth K, Bourke MJ. Deep mural injury and perforation after colonic endoscopic mucosal resection: a new classification and analysis of risk factors. Gut. 2017 Oct;66(10):1779-1789. doi: 10.1136/gutjnl-2015-309848. Epub 2016 Jul 27. PMID 27464708